CLINICAL TRIAL: NCT03397095
Title: Sequential Treatment of Extra-Corporeal Shock Wave Combined With aUtologous Bone marRow Mesenchymal Stem Cells in Patients With ischEmic Heart Disease : the S-CURE Study
Brief Title: Sequential Treatment of Extra-Corporeal Shock Wave Combined With aUtologous Bone marRow Mesenchymal Stem Cells on Patients With ischEmic Heart Disease : the S-CURE Study
Acronym: S-CURE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-CURE
Record Dates: First submitted 2017-12-28; First posted 2018-01-11 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Ischemic Heart Disease
Keywords: stem cells, ischemic heart disease.
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: S-CURE study has a two-stage design. Stage 1 is an open-labled, lead-in study. 20 participants will be enrolled in this stage. It is conducted to assess the feasibility and safety of the study procedures as well as the bioactivity of the products. Stage 2 is an randomized, placebo controlled study, 100 participants will be enrolled in this stage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSWT+BMMSCs (Experimental): Patients in CSWT+BMMSCs group will receive a 3-month cardiac shock wave therapy and then a total of 1 million/kg BMMSCs will be infused using the stop-flow technique through an over-the-wire balloon catheter positioned in a coronary artery or bypass graft supplying the targeting viable myocardium.
  Interventions: Combination Product: CSWT+BMMSCs
- CSWT+Sham operation (Sham Comparator): Placebo group will receive a 3-month CSWT and a sham procedure.
  Interventions: Device: CSWT+Sham operation

INTERVENTIONS:
Combination Product: CSWT+BMMSCs — All participants will screened by D-SPECT to assess the myocardium viability. If the viable myocardium is detected, Patients will be randomized to receive cardiac shock wave therapy with an equipment (Modulith SLC; Storz Medical, Switzerland) followed the recommended protocol developed by Tohoku University of Japan and the protocol developed by the University of Essen, Germany. An over-the-wire catheter will be positioned in the target coronary artery and the cells resuspended in saline will be injected intracoronary.
  Arms: CSWT+BMMSCs
Device: CSWT+Sham operation — Patients randomized to this group will receive a routine cardiac shock wave therapy and coronary angiography. No cells will be administered via the coronary artery.
  Arms: CSWT+Sham operation

SUMMARY:
This study is designed to evaluate the efficacy, safety and tolerability of autologous bone marrow derived mesenchymal stem cells compared to placebo (sham operation) when administered via percutaneous coronary infusion to patients with ischemic heart disease, who are screened by D-SPECT and have pretreated with 3-month cardiac shock wave therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females;
2. Chronic ischemic heart failure, previous anterior myocardial infarction > 3months;
3. Viable myocardium is detected by D-SPECT;
4. LVEF < 50% measured by echocardiography or NYHA II-IV;
5. No planed reasonable revascularization procedures;
6. At least 30 days standard medical therapy for heart failure before screening;
7. Worsening heart failure within 6 months or have a NT-proBNP ≥1000 pg/mL or BNP ≥200 pg/mL within 30 days of screening (including screening); or have a 6-minute walk test (6MWT) distance of ≤425 meters at screening;
8. Written informed consent.

Exclusion Criteria:

1. Ventricular thrombus;
2. Myocardial infarction, TIA or stroke < 3 months;
3. CRT/CRT-D implantation, heart transplantation, cardiomyoplasty, left ventricular reduction surgery, heart failure-related device interventions, or cardiac shunt implantation;
4. Active infection or fever;
5. Chronic inflammatory disease;
6. HIV infection or active hepatitis;
7. Hemoglobin A1c (HbA1c) ≥ 9% at screening;
8. Body mass index (BMI) ≥ 40 kg/m2 at screening;
9. Chronic kidney disease (CKD) requiring dialysis (Stage 5) or estimated creatinine clearance < 30 mL/min/1.73㎡ at screening;
10. Allergies to any equine, porcine, or bovine products;
11. Abnormal laboratory values at screening：Platelets < 50,000 μL;Hemoglobin < 9.0 g/dL; Aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 3 times the upper limit of normal (ULN);
12. Pregnancy;
13. Mental retardation;
14. Participation in other clinical study < 1 month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months follow-up in LVEF. | 6 months
  The primary outcome will evaluate the change in left ventricular function as measured by echocardiography and D-SPECT for left ventricular ejection fraction (LVEF).
Change from baseline to 6 months follow-up in infarct size. | 6 months
  The primary outcome will evaluate the change in infarct size as measured by D-SPECT.

SECONDARY OUTCOMES:
Change from baseline to 6 months follow-up in exercise distance increment | 6 months
  A secondary objective will be the changes from baseline to 6 months post-treatment in the distance walked as measured by the 6-minute walk test.
Change from baseline to 6 months follow-up in quality of life measured by MLHFQ | 6 months
  A secondary objective will be the change in quality of life in patients treated with bone marrow derived mesenchymal stem cells compared to placebo using the Minnesota Living with Heart Failure Questionnaire (MLHFQ).
Change from baseline to 6 months follow-up in NYHA Classification. | 6 months
  A secondary objective will be the change from baseline to Month 6 in NYHA Classification in patients treated with BMMSCs compared to placebo.
Percent of patients with adverse events. | 6 months
  A secondary objective will be the overall safety and tolerability of BMMSCs versus placebo in patients with ICM from time of cell-infusion through 6 months post-treatment follow-up by the percentage of patients with adverse events.
Change from baseline to 6 months follow-up in exercise time increment. | 6 months
  A secondary objective will be the changes from baseline to 6 months post-treatment in the exercise time as measured by the cardiopulmonary exercise test.
Change from baseline to 6 months follow-up in quality of life measured by KCCQ | 6 months
  A secondary objective will be the change in quality of life in patients treated with bone marrow derived mesenchymal stem cells compared to placebo using the Kansas City Cardiomyopathy Questionnaire (KCCQ).

OTHER OUTCOMES:
Percent of patients with major adverse cardiac events (MACE) | 6 months
  A secondary objective will be the overall safety and tolerability of BMMSCs versus placebo in patients with ICM by the percentage of patients who experience MACE events. MACE events include: unstable angina requiring hospitalization, myocardial infarction, stroke, worsening heart failure requiring hospitalization, VAD implantation, heart transplant, resuscitated sudden death, and cardiovascular death.
Average number of clinical events over 12 months post-treatment | 12 months
  A secondary outcome will assess the efficacy of BMMSc compared to placebo on the average number of events per patient over 12 months post-treatment in each treatment arm (total number events in each arm/total number of patients in each arm). The events include: all-cause deaths, cardiovascular hospitalizations, and unplanned outpatient or emergency department visits to treat acute decompensated heart failure. The clinical events used in this endpoint will be adjudicated by an independent clinical endpoint committee who are blinded to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD,PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Intracoronary bone marrow-derived progenitor cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1210-21. doi: 10.1056/NEJMoa060186. PMID 16990384
- [Background] Assmus B, Walter DH, Seeger FH, Leistner DM, Steiner J, Ziegler I, Lutz A, Khaled W, Klotsche J, Tonn T, Dimmeler S, Zeiher AM. Effect of shock wave-facilitated intracoronary cell therapy on LVEF in patients with chronic heart failure: the CELLWAVE randomized clinical trial. JAMA. 2013 Apr 17;309(15):1622-31. doi: 10.1001/jama.2013.3527. PMID 23592107
- [Background] Patel AN, Henry TD, Quyyumi AA, Schaer GL, Anderson RD, Toma C, East C, Remmers AE, Goodrich J, Desai AS, Recker D, DeMaria A; ixCELL-DCM Investigators. Ixmyelocel-T for patients with ischaemic heart failure: a prospective randomised double-blind trial. Lancet. 2016 Jun 11;387(10036):2412-21. doi: 10.1016/S0140-6736(16)30137-4. Epub 2016 Apr 5. PMID 27059887
- [Background] Bonow RO, Maurer G, Lee KL, Holly TA, Binkley PF, Desvigne-Nickens P, Drozdz J, Farsky PS, Feldman AM, Doenst T, Michler RE, Berman DS, Nicolau JC, Pellikka PA, Wrobel K, Alotti N, Asch FM, Favaloro LE, She L, Velazquez EJ, Jones RH, Panza JA; STICH Trial Investigators. Myocardial viability and survival in ischemic left ventricular dysfunction. N Engl J Med. 2011 Apr 28;364(17):1617-25. doi: 10.1056/NEJMoa1100358. Epub 2011 Apr 4. PMID 21463153